CLINICAL TRIAL: NCT06053853
Title: Safety Profile of Diphtheria Antitoxin (DAT) in Indonesia
Brief Title: Post Marketing Surveillance of Diphtheria Antitoxin (DAT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAT 0422
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Safety Issues
MeSH Terms: interventions — Diphtheria Antitoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Product (Experimental): Diphtheria Antitoxin (DAT)
  Administered intravenously.
  Dosage:
  * Mild diphtheria (nose, skin): 20,000 unit
  * Moderate diphtheria (tonsil - limited): 40,000 - 60,000 unit
  * Severe diphtheria (more than 1 tonsil, or to the pharyngeal wall, or more than 5 days of illness, or with bull neck): 80,000 - 120,000 unit
  Interventions: Biological: Diphtheria Antitoxin

INTERVENTIONS:
Biological: Diphtheria Antitoxin — Dosage form: Solution for injection
  Dosage:
  1. Perform sensitivity tests, and desensitization if necessary.
  2. Give the entire treatment dose of antitoxin IV (or IM) in a single administration (except for series of injections needed for desensitization).
  3. The recommended DAT treatment dosage ranges (pediatric and adult) are:
     * Pharyngeal or laryngeal disease of 2 days duration 20,000 - 40,000 unit
     * Nasopharyngeal disease 40,000 - 60,000 unit
     * Extensive disease of 3 or more days duration, or any patient with diffuse swelling of neck 80,000 - 100,000 unit
     * Skin lesions only (rare case where treatment is indicated) 20,000 - 40,000 unit

SUMMARY:
The aim of this study is to evaluate the safety profile of Diphtheria Antitoxin

DETAILED DESCRIPTION:
To assess the occurrence of serum sickness after Diphtheria Antitoxin administration.

To assess local and systemic reactions within 24 hours to 10 days. To assess the occurrence of positive reactions after the sensitivity test (skin test). To assess the presence of SAE after Diphtheria Antitoxin administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a probable diagnosis or laboratory confirmation of Diphtheria.
* Subjects who received therapy with the intended DAT

Exclusion Criteria:

* Receiving a different brand of Diphtheria Antitoxin (DAT)

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
The occurrence of serum sickness after administration of Diphtheria Antitoxin (DAT) | Within 10 days after injection
  Percentage of serum sickness after administration of Diphtheria Antitoxin (DAT)

SECONDARY OUTCOMES:
The occurrence of local and systemic reactions after administration of Diphtheria Antitoxin (DAT) | Within 24 hours to 10 days after injection
  Percentage of local and systemic reaction after administration of Diphtheria Antitoxin (DAT)
The occurrence of positive reaction after a sensitivity test (skin test) of Diphtheria Antitoxin (DAT) | Before injection of Diphtheria Antitoxin
  Percentage of positive reaction after sensitivity test (skin test) of Diphtheria Antitoxin (DAT)
The occurrence of serious adverse event (SAE) after administration of Diphtheria Antitoxin (DAT) | Within 10 days after injection
  Percentage of serious adverse event (SAE) after administration of Diphtheria Antitoxin (DAT)

CONTACTS AND LOCATIONS:
Overall Officials: Dominicus Husada, MD, Principal Investigator — Dr. Soetomo Hospital, Surabaya, Indonesia
Locations (1):
- RSUD Dr. Soetomo, Surabaya, East Java, Indonesia